CLINICAL TRIAL: NCT06646757
Title: Exploring Multiple Self-Help Interventions to Promote Self-Efficacy and Overcome Disability
Acronym: EMPOWER-IBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 853060
Record Dates: First submitted 2024-08-21; First posted 2024-10-17 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Ulcerative Colitis (UC); Crohn Disease (CD)
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Arm 1 (No Intervention): No resource provision
- Arm 2 (Experimental): Power of Two (PEER) is a one-on-one peer mentoring program operated by the Crohn's & Colitis Foundation
  Interventions: Behavioral: PEER
- Arm 3 (Experimental): IBD Help Center (HELP) is a resource operated by the Crohn's and Colitis Foundation (CCF) for individuals to connect with an information specialist via email, call, or online live chat at no cost
  Interventions: Behavioral: HELP
- Arm 4 (Experimental): IBD Help Center (HELP) is a resource operated by the Crohn's and Colitis Foundation (CCF) for individuals to connect with an information specialist via email, call, or online live chat at no cost Power of Two (PEER) is a one-on-one peer mentoring program operated by the Crohn's & Colitis Foundation
  Interventions: Behavioral: HELP; Behavioral: PEER
- Arm 5 (Experimental): "Coping with Crohn's and Colitis: A Patient and Clinician's Guide to CBT for IBD" (CBT) is an IBD-specific cognitive behavioral therapy (CBT) workbook (e-book or hardcopy)
  Interventions: Behavioral: CBT
- Arm 6 (Experimental): "Coping with Crohn's and Colitis: A Patient and Clinician's Guide to CBT for IBD" (CBT) is an IBD-specific cognitive behavioral therapy (CBT) workbook (e-book or hardcopy)
  Power of Two (PEER) is a one-on-one peer mentoring program operated by the Crohn's & Colitis Foundation
  Interventions: Behavioral: CBT; Behavioral: PEER
- Arm 7 (Experimental): "Coping with Crohn's and Colitis: A Patient and Clinician's Guide to CBT for IBD" (CBT) is an IBD-specific cognitive behavioral therapy (CBT) workbook (e-book or hardcopy) IBD Help Center (HELP) is a resource operated by the Crohn's and Colitis Foundation (CCF) for individuals to connect with an information specialist via email, call, or online live chat at no cost
  Interventions: Behavioral: CBT; Behavioral: HELP
- Arm 8 (Experimental): "Coping with Crohn's and Colitis: A Patient and Clinician's Guide to CBT for IBD" (CBT) is an IBD-specific cognitive behavioral therapy (CBT) workbook (e-book or hardcopy) IBD Help Center (HELP) is a resource operated by the Crohn's and Colitis Foundation (CCF) for individuals to connect with an information specialist via email, call, or online live chat at no cost Power of Two (PEER) is a one-on-one peer mentoring program operated by the Crohn's & Colitis Foundation
  Interventions: Behavioral: CBT; Behavioral: HELP; Behavioral: PEER
- Arm 9 (Experimental): 1) My IBD Care (APP) is a free smartapp that supports patients' tracking of symptoms, medical appointments, and medications; self-paced behavioral change programs
  Interventions: Behavioral: APP
- Arm 10 (Experimental): My IBD Care (APP) is a free smartapp that supports patients' tracking of symptoms, medical appointments, and medications; self-paced behavioral change programs
  Power of Two (PEER) is a one-on-one peer mentoring program operated by the Crohn's & Colitis Foundation
  Interventions: Behavioral: APP; Behavioral: PEER
- Arm 11 (Experimental): My IBD Care (APP) is a free smartapp that supports patients' tracking of symptoms, medical appointments, and medications; self-paced behavioral change programs
  IBD Help Center (HELP) is a resource operated by the Crohn's and Colitis Foundation (CCF) for individuals to connect with an information specialist via email, call, or online live chat at no cost
  Interventions: Behavioral: APP; Behavioral: HELP
- Arm 12 (Experimental): My IBD Care (APP) is a free smartapp that supports patients' tracking of symptoms, medical appointments, and medications; self-paced behavioral change programs
  IBD Help Center (HELP) is a resource operated by the Crohn's and Colitis Foundation (CCF) for individuals to connect with an information specialist via email, call, or online live chat at no cost
  Power of Two (PEER) is a one-on-one peer mentoring program operated by the Crohn's & Colitis Foundation
  Interventions: Behavioral: APP; Behavioral: HELP; Behavioral: PEER
- Arm 13 (Experimental): My IBD Care (APP) is a free smartapp that supports patients' tracking of symptoms, medical appointments, and medications; self-paced behavioral change programs
  "Coping with Crohn's and Colitis: A Patient and Clinician's Guide to CBT for IBD" (CBT) is an IBD-specific cognitive behavioral therapy (CBT) workbook (e-book or hardcopy)
  Interventions: Behavioral: APP; Behavioral: CBT
- Arm 14 (Experimental): My IBD Care (APP) is a free smartapp that supports patients' tracking of symptoms, medical appointments, and medications; self-paced behavioral change programs
  "Coping with Crohn's and Colitis: A Patient and Clinician's Guide to CBT for IBD" (CBT) is an IBD-specific cognitive behavioral therapy (CBT) workbook (e-book or hardcopy)
  Power of Two (PEER) is a one-on-one peer mentoring program operated by the Crohn's & Colitis Foundation
  Interventions: Behavioral: APP; Behavioral: CBT; Behavioral: PEER
- Arm 15 (Experimental): My IBD Care (APP) is a free smartapp that supports patients' tracking of symptoms, medical appointments, and medications; self-paced behavioral change programs
  "Coping with Crohn's and Colitis: A Patient and Clinician's Guide to CBT for IBD" (CBT) is an IBD-specific cognitive behavioral therapy (CBT) workbook (e-book or hardcopy)
  IBD Help Center (HELP) is a resource operated by the Crohn's and Colitis Foundation (CCF) for individuals to connect with an information specialist via email, call, or online live chat at no cost
  Interventions: Behavioral: APP; Behavioral: CBT; Behavioral: HELP
- Arm 16 (Experimental): 1. My IBD Care (APP) is a free smartapp that supports patients' tracking of symptoms, medical appointments, and medications; self-paced behavioral change programs
  2. "Coping with Crohn's and Colitis: A Patient and Clinician's Guide to CBT for IBD" (CBT) is an IBD-specific cognitive behavioral therapy (CBT) workbook (e-book or hardcopy)
  3. IBD Help Center (HELP) is a resource operated by the Crohn's and Colitis Foundation (CCF) for individuals to connect with an information specialist via email, call, or online live chat at no cost
  4. Power of Two (PEER) is a one-on-one peer mentoring program operated by the Crohn's & Colitis Foundation
  Interventions: Behavioral: APP; Behavioral: CBT; Behavioral: HELP; Behavioral: PEER

INTERVENTIONS:
Behavioral: APP — 1) My IBD Care (APP) is a free smartapp that supports patients' tracking of symptoms, medical appointments, and medications; self-paced behavioral change programs
  Arms: Arm 10; Arm 11; Arm 12; Arm 13; Arm 14; Arm 15; Arm 16; Arm 9
Behavioral: CBT — 2) "Coping with Crohn's and Colitis: A Patient and Clinician's Guide to CBT for IBD" (CBT) is an IBD-specific cognitive behavioral therapy (CBT) workbook (e-book or hardcopy)
  Arms: Arm 13; Arm 14; Arm 15; Arm 16; Arm 5; Arm 6; Arm 7; Arm 8
Behavioral: HELP — 3) IBD Help Center (HELP) is a resource operated by the Crohn's and Colitis Foundation (CCF) for individuals to connect with an information specialist via email, call, or online live chat at no cost
  Arms: Arm 11; Arm 12; Arm 15; Arm 16; Arm 3; Arm 4; Arm 7; Arm 8
Behavioral: PEER — 4) Power of Two (PEER) is a one-on-one peer mentoring program operated by the Crohn's & Colitis Foundation
  Arms: Arm 10; Arm 12; Arm 14; Arm 16; Arm 2; Arm 4; Arm 6; Arm 8

SUMMARY:
EMPOWER-IBD aims to identify behavioral interventions to strengthen patients' self-efficacy for self-management as a mechanism to reduce IBD-related disability. This multisite, randomized controlled trial with 16 arms will randomize adults with moderate-to-severe IBD-related disability to a combination of four multimodal behavioral interventions to test their clinical effectiveness in reducing IBD-related disability and improving self-efficacy. The interventions are four existing, publicly available disease-specific self-help resources offered at no cost to the participants: a book, smart app, help center, and peer mentor. Participants will complete online surveys and may engage in virtual focus groups. Participants may receive an honorarium (e-gift card) and/or be entered into a lottery for a giftcards post-survey completion and focus group participation.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (age ≥ 18 years) with IBD and moderate-to-severe IBD-related (IBD) Disability Index score > 35 26,27)
2. Able to consent, complete surveys, and participate in focus groups in English.

Exclusion Criteria:

1. No/low disability (IBD-DI < 35) on the baseline survey
2. Inability or unwillingness to participate in the interventions
3. Inability to download apps from the Apple AppStore or Google Play store (necessary to engage with the smartapp intervention)
4. Limited English proficiency (necessary because some interventions are currently only offered in English)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 803 (Actual)
Dates: Start 2024-08-14 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Change in IBD-related disability based on the validated IBD-Disability Index | 12 weeks
  The study seeks to identify any changes in IBD-related disability pre-post intervention (week 0 and week 12) as measured by the IBD Disability Index (IBD-DI). IBD-related disability is measured by the validated 14-item IBD-disability index (yes-no responses and 1-5 point Likert scales) for limitations across 5 domains of International Classification of Functioning, Health, and Disability. Higher score indicates more disability. Total score ranges from 0-100, interpreted as 0-20 (no disability), 20-35 (mild disability), 35-50 (moderate disability), and 50-100 (severe disability).

SECONDARY OUTCOMES:
Change in IBD self-efficacy as measured by the IBD Self-Efficacy Scale Wasson Health Confidence Scale | 12 weeks
  The study seeks to identify any changes in IBD self-efficacy as measured in the 13-item IBD-Self Efficacy Wasson Health Confidence Scale. This is one survey. A higher score indicates more confidence in self-efficacy and health confidence relative to chronic illness. Total score ranges from 0-130

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No